CLINICAL TRIAL: NCT00252135
Title: An Epidemiologic Study of Xolair (Omalizumab): Evaluating Clinical Effectiveness and Long-Term Safety in Patients With Moderate to Severe Asthma (EXCELS)
Brief Title: A Study of Xolair to Evaluate Effectiveness and Long-Term Safety in Patients With Moderate to Severe Asthma
Status: Completed | Type: Observational
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Q2948g
Record Dates: First submitted 2005-11-09; First posted 2005-11-11 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Asthma
Keywords: Moderate to severe asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study is a multicenter, prospective, observational cohort study of ~5000 Xolair-treated and ~2500 non-Xolair-treated patients with moderate to severe persistent asthma and a positive skin test or in vitro reactivity to an aeroallergen.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent document (in the case of a minor, consent must be given by the child's parent or legally authorized representative)
* ≥12 years of age
* Physician diagnosis of moderate to severe persistent asthma
* Evidence or history of positive skin test or in vitro reactivity to an aeroallergen
* Willingness to participate fully for the duration of the study (5 years)
* For patients in the Xolair-treated cohort, have received at least one dose of Xolair therapy at the time of enrollment

Exclusion Criteria:

* Contraindication to Xolair therapy (e.g., patients who experienced a severe hypersensitivity reaction to Xolair)
* Acute asthma exacerbation within the previous 2 weeks of screening requiring any of the following: initiation of systemic corticosteroids, increased doses of systemic corticosteroids from baseline, doubling of inhaled corticosteroids, emergency room visit, or hospitalization
* Acute flare of significant systemic disease (e.g., infection, hematologic, renal, hepatic, cardiovascular diseases, or gastrointestinal diseases), or a recent hospitalization because of their disease within the previous 2 months
* Use of an experimental drug within 30 days prior to study screening
* Diagnosis of cystic fibrosis
* For patients in the non-Xolair-treated cohort, any prior treatment with Xolair

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be recruited from a variety of practice settings, including managed care organizations, community physicians, and academic centers.
Sampling Method: Non-Probability Sample
Enrollment: 8023 (Actual)
Dates: Start 2004-06 (Actual); Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Wong, M.D., Study Director — Genentech, Inc.

REFERENCES:
- [Derived] Fiocchi A, Chinthrajah RS, Ansotegui IJ, Sriaroon P, Mustafa SS, Raut P, Cameron B, Gupta S, Fleischer DM. Does Comorbid Food Allergy Affect Response to Omalizumab in Patients with Asthma? J Asthma Allergy. 2024 Sep 17;17:889-900. doi: 10.2147/JAA.S475517. eCollection 2024. PMID 39309477
- [Derived] Eisner MD, Yegin A, Trzaskoma B. Severity of asthma score predicts clinical outcomes in patients with moderate to severe persistent asthma. Chest. 2012 Jan;141(1):58-65. doi: 10.1378/chest.11-0020. Epub 2011 Sep 1. PMID 21885725
- [Derived] Long AA, Fish JE, Rahmaoui A, Miller MK, Bradley MS, Taki HN, Demeo AN, Tilles SA, Szefler SJ. Baseline characteristics of patients enrolled in EXCELS: a cohort study. Ann Allergy Asthma Immunol. 2009 Sep;103(3):212-9. doi: 10.1016/S1081-1206(10)60184-6. PMID 19788018
- [Derived] Wechsler ME, Wong DA, Miller MK, Lawrence-Miyasaki L. Churg-strauss syndrome in patients treated with omalizumab. Chest. 2009 Aug;136(2):507-518. doi: 10.1378/chest.08-2990. Epub 2009 May 1. PMID 19411292